CLINICAL TRIAL: NCT03573219
Title: A New Experimental Model of Acute Muscle Pain in Humans Based on Short-wave Diathermy
Brief Title: A New Experimental Model of Transient and Short-lasting Muscle Pain in Humans Based on Diathermy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, José Biurrun Manresa, Principal Investigator, National Council of Scientific and Technical Research, Argentina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IS001890
Record Dates: First submitted 2018-06-05; First posted 2018-06-29 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Injury
Keywords: Short-Wave Diathermy; Transient muscle pain; Non-invasive pain model
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: The SWD applicators will be placed in the desired position, around the forearm for the upper limb experiments, or below the knee for the lower limb experiments. The distance between applicators will be adjusted until the desired pain sensation is obtained according to the subjective criterion of the volunteer. This sensation should be mild or moderate pain, but tolerable for the duration of the application. Once the first application is completed, the volunteer will be allowed to rest for a period of 10 minutes, and the assessment will be repeated to test for possible after effects. After it is verified that the muscles recovered their normal temperature and the pain sensation has completely disappeared, the variables related to changes in motor responses under rest conditions will be recorded. Then SWD will be applied a second time using the same parameters as in the first application. Once the registration is complete, the experiment will be finished.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy participant (Experimental): Healthy volunteers that fulfill the inclusion criteria. Intervention: Short-wave diathermy (Radiation)
  Interventions: Radiation: Short-wave diathermy

INTERVENTIONS:
Radiation: Short-wave diathermy — The application of SWD will be carried out by a CEC M-8 short-wave thermotherapy unit. The device has capacitive applicators, that will be situated around the muscle to be irradiated on top of a cotton towel, in order to absorb perspiration and avoid undesired heating effects. Afterwards the emission mode (continuous or pulsed) will be selected, and application of SWD will start. The intensity of SWD will be gradually increased until the volunteer perceives a warm sensation, and once familiarized with this perception, the intensity will be increased until a sensation of constant but tolerable pain is evoked. This sensation will be maintained throughout the duration of the SWD application, estimated in approximately 10 minutes.

SUMMARY:
This study evaluates the use of short-wave diathermy (SWD) as an novel experimental model to induce transient and intensity-controlled muscle pain by heating muscle tissue.

DETAILED DESCRIPTION:
Application of short-wave diathermy All researchers, students and postdocs involved in experimental application of SWD will be properly trained by the Non-Ionizing Radiation Research Group of the National University of Entre Ríos. The application of SWD will be carried out by a CEC M-8 short-wave thermotherapy unit (CEC Electrónica, Córdoba, Argentina). The device has capacitive applicators, that will be situated around the muscle to be irradiated on top of a cotton towel, in order to absorb perspiration and avoid undesired heating effects. Afterwards the emission mode (continuous or pulsed) will be selected, and application of SWD will start. The intensity of SWD will be gradually increased until the volunteer perceives a warm sensation, and once familiarized with this perception, the intensity will be increased until a sensation of constant but tolerable pain is evoked. This sensation will be maintained throughout the duration of the SWD application, estimated in approximately 10 minutes. In case the volunteer feels excessive discomfort or does not adequately tolerate the application of SWD, the device will be turned off immediately and the experimental session will finish.

Experimental pain model assessment

* Model direct effects: maximum and average pain ratings will be assessed through a Visual Analog Scale (VAS). The VAS ranges from 0 to 10, where 0 represents no perception, 3 represents the pain threshold (i.e. the minimum irradiation intensity that elicits pain) and 10 represents the tolerance threshold (i.e. the irradiation intensity that elicits an intolerable pain sensation). Duration of pain will also be recorded, in case the experiment has to be interrupted before SWD application is completed and to assess potential cases in which pain outlasts SWD application. Furthermore, delivered RF power will be measured using a Bird 43 RF wattmeter (Bird Technologies, OH, USA).
* Pressure stimulation: pressure stimulation will be applied through a Somedic algometer (Somedic SenseLab AB, Sweden), directly over the muscle being examined, using a 1 cm2 round tip. Pressure will be gradually increased from 0 kPA until a maximum of 1000 kPa at a rate of approximately 30 kPa/s. Pressure pain threshold (PPT) will be defined as the force at which the pressure sensation becomes painful. Pressure tolerance threshold (PTT) will be defined as the force at which pressure sensation becomes intolerable. If any of the threshold are not reached until the pressure is increased to 1000 kPa, the this value will be considered as the corresponding threshold.
* Pinprick and tactile stimulation: pinprick stimuli will be applied on the skin over the muscle being examined using a set of pinprick stimulators, consisting on a needle with a 0.25 mm tip linked to calibrated weights, ranging from 1 g to 50 g, in order to apply forces between 8 and 500 mN approximately. Dynamic tactile stimulation will be applied by stroking a cotton tip over the skin. Pinprick sensitivity (PS) and dynamic tactile sensitivity (DTS) will be quantified using the VAS described above.
* Electrical stimulation: electrical stimuli will be applied to the skin over the muscle being examined using a concentric electrode, in which the cathode is made of 16 stainless steel blunt pins with 0.2 mm diameter tips and 1 mm length, and the anode is a concentric stainless steel ring of 20 mm diameter. The electrical stimulus will consist on a rectangular pulse of 1 ms duration, generated by a Biopac STMISOLA constant-current electrical stimulator (Biopac Systems Inc., California, USA). Stimulation intensity will be increased from 1 mA in steps of 0.5 mA until a pain sensation is evoked. This intensity will be defined as the electrical pain threshold (EPT). Once the EPT is determined, repeated stimulation will be applied referenced to this intensity in order to record somatosensory evoked potentials (SEPs) through surface electroencephalography (EEG).
* Motor responses: motor responses will be recorded from upper and lower limbs. For the upper limb, two sets of experimental motor tasks are planned, and the overall aim is to measure changes in precision in the execution of the motor tasks due to pain. The first one will be a simple task, basically consisting on the use of a joystick to move a cursor to a two-dimensional moving target displayed in a computer screen. Specific details of the implementation of the optimal setup for this motor task and the required software will be provided by collaborators from the Physiology of Action Lab at Universidad de Buenos Aires. The second motor task will involve more complex movements and haptic feedback, provided by a Phantom Omni haptic device (SensAble Technologies, Inc., Massachusetts, USA). The haptic device can provide controlled levels of force feedback (up to 3.3 N) and a precise mapping of the trajectories employed in the motor task in three dimensions (resolution: 0.055 mm). Specific details of the implementation of the optimal setup for this motor task and the required software will be provided by collaborators from the Robotics Research Group at National University of Entre Ríos. For the lower limb, the motor task will consist on a balance task performed over high-resolution pressure sensing platform that will be able to record differences in weight loading between left and right leg and variations in the center of pressure (CoP). The platform is a recent technological development from the Electronic Prototyping and 3D Printing Lab at the Faculty of Engineering of National University of Entre Ríos, and it has a sensing area of 430 x 320 mm, with a resolution of 4 pressure sensors per cm2 and a measurement range from 1 to 785 kPa.
* Brain responses: EEG will be recorded using a Neuroscan SynAmps amplifier (Compumedics Ltd., Victoria, Australia) during the planning and execution of motor tasks, in order to evaluate changes in movement-related cortical potentials (MRCP) in relation to SWD-induced pain (Jochumsen et al. 2015). Additionally, resting-state EEG will be recorded before, during and after SWD application, in order to assess potential changes in functional connectivity (FC) (Mayhew et al. 2013). FC analysis will be performed by collaborators from CNAP at Aalborg University.

Sample size considerations

The experimental design is an interventional, pre-post study design (Thiese 2014), in which each participant acts as his own control. Sample size calculation will be performed taking into account the expected effect size that the model will have on the primary outcome (PPT). Several experiments have shown that PPT in the wrist extensor/flexor muscles (e.g. extensor carpi radialis longus) is around 350 ± 150 kPa (mean ± standard deviation), whereas PPT for the ankle dorsiflexor muscles (e.g. tibialis anterior) is around 600 ± 250 kPa (Fischer 1987; Delfa de la Morena et al. 2013). On the other hand, there is no existing information on the expected size of the difference in PPT due to the application of SWD, so this value will be approximated taking into account reference values of differences in PPT generated by other experimental models of pain, such as the injection of hypertonic saline solution or delayed onset muscle soreness. In these cases, PPT is usually reduced between 10 and 30% during the effects of the model, so an average of 20% difference will be considered in order to calculate the sample size for these experiments. Considering a probability of making a type I error (α) of 5%, a statistical power (1 - β) of 80%, and an estimated correlation between measures of 0.8, the sample size required to detect the aforementioned difference is 16 volunteers for the experiment in the upper limb and 17 volunteers for the experiment in the lower limb. In order to account for an unexpectedly larger variation, 20 subjects are expected to be recruited for each experiment.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the content and scope of the experiment, and compliance with the experiment's instructions.
* To have signed the informed consent.

Exclusion Criteria:

* Pregnancy.
* Previous history of neurological or musculoskeletal disorders or chronic pain.
* Previous history of addictive behavior, defined as abuse of alcohol, cannabis, opioids or other drugs.
* Previous history of thermosensitivity disorders.
* Previous history of mental illness.
* Presence of fever, tuberculosis, tumors, infectious processes, or acute inflammatory processes.
* Implantation of peacemaker or metallic prosthesis.
* Use of analgesics within 24 h prior to the experiment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) | 0 to 1 hour
  Change in the pressure pain threshold (kPa) recorded after the induced of muscle pain using SWD on the established time point records.

SECONDARY OUTCOMES:
Assessment of changes in pain intensity in direct relation to the experimental model | 0 to 1 hour
  Maximum and average pain ratings (0 to 100 score).
Assessment of changes in pain time course in direct relation to the experimental model | 0 to 1 hour
  Duration of pain (seconds)
Assessment of changes in functional connectivity in direct relation to the experimental model | 0 to 1 hour
  Changes in functional connectivity (FC), assessed through surface electroencephalography (EEG).
Assessment of changes in Pinprick sensitivity | 0 to 1 hour
  Pinprick sensitivity (PS) (0 to 100 score).
Assessment of changes in Dynamic tactile sensitivity | 0 to 1 hour
  Dynamic tactile sensitivity (DTS) (0 to 100 score).
Assessment of changes in Electrical pain threshold | 0 to 1 hour
  Electrical pain threshold (EPT) (mA).
Assessment of changes in Somatosensory evoked potentials | 0 to 1 hour
  Somatosensory evoked potentials in response to electrical stimuli (SEP), assessed through EEG. (mV)
Assessment of changes in Movement-related cortical potentials | 0 to 1 hour
  Change in Movement-related cortical potentials (MRCP), assessed through EEG.
Assessment of changes in motor responses for upper limb | 0 to 1 hour
  Change in precision during motor execution (percentage)
Assessment of changes in motor responses for lower limb | 0 to 1 hour
  Change in balance (Centre of pressure)
Assessment of changes in weight loading | 0 to 1 hour
  Measured in Kg

CONTACTS AND LOCATIONS:
Overall Officials: José Biurrun Manresa, PhD, Principal Investigator — National Scientific and Technical Research Council - Argentina
Locations (1):
- Facultad de Ingeniería - Universidad Nacional de Entre Ríos (Argentina), Oro Verde, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From first date of publication of journal article.
Access Criteria: IPD will be provided upon request.

REFERENCES:
- [Background] Goats GC. Continuous short-wave (radio-frequency) diathermy. Br J Sports Med. 1989 Jun;23(2):123-7. doi: 10.1136/bjsm.23.2.123. PMID 2691003
- [Background] Graven-Nielsen T. Fundamentals of muscle pain, referred pain, and deep tissue hyperalgesia. Scand J Rheumatol Suppl. 2006;122:1-43. doi: 10.1080/03009740600865980. No abstract available. PMID 16997767
- [Background] Neziri AY, Scaramozzino P, Andersen OK, Dickenson AH, Arendt-Nielsen L, Curatolo M. Reference values of mechanical and thermal pain tests in a pain-free population. Eur J Pain. 2011 Apr;15(4):376-83. doi: 10.1016/j.ejpain.2010.08.011. Epub 2010 Oct 6. PMID 20932788
- [Background] Vuilleumier PH, Biurrun Manresa JA, Ghamri Y, Mlekusch S, Siegenthaler A, Arendt-Nielsen L, Curatolo M. Reliability of Quantitative Sensory Tests in a Low Back Pain Population. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):665-73. doi: 10.1097/AAP.0000000000000289. PMID 26222349